CLINICAL TRIAL: NCT02334774
Title: Effects of an Swallowing and Oral Care Program on Swallowing and Oral Intake Status in Patients Following Prolonged Endotracheal Intubation
Brief Title: Effects of an Swallowing and Oral Care Program in Patients Following Prolonged Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201411079RIND
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2016-04

CONDITIONS: Dysphagia; Endotracheal Intubation; Intake Status; Swallowing Status
MeSH Terms: conditions — Deglutition Disorders | interventions — Deglutition

STUDY DESIGN:
Intervention Model Description: Pre-and post- intervention
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants receiving an SOC Program (Experimental): Participants following prolonged endotracheal intubation receiving a up to 14-day daily Swallowing and Oral Care Program.
  Interventions: Procedure: Swallowing and Oral Care Program

INTERVENTIONS:
Procedure: Swallowing and Oral Care Program — An Swallowing and Oral Care Program involves moisturizing and cleansing oral cavity, massaging salivary gland, oral motor exercise daily, and intake education as needed.

SUMMARY:
This pre-and post-intervention study enrolled adult Intensive Care Unit(ICU) patients (≥50 years) successfully extubated after ≥48 hours endotracheal intubation and without preexisting neuromuscular disease or swallowing dysfunction.

All participants received by a trained nurse-administered, hospital-based (up to 14 days) Swallowing and Oral Care(SOC) intervention comprising toothbrushing/salivary gland massage, oral motor exercise, and advice on safe-swallowing strategies.

All participants' daily intake status (21 days) and oral health status, oral sensation(stereognosis, light touch and two-point discrimination), tongue and lip strength, salivary secretion, body weight) were assessed at 2, 7, 14 days post-extubation by a blinded research nurse.

Feasibility was evaluated as time spent providing SOC, patients adherence to SOC components, and adverse event(i.e., coughing, wet voice, or decreased oxygen saturation) during SOC intervention.

DETAILED DESCRIPTION:
With rapid growth of medical technology, patients receiving oral endotracheal intubation have increased. Although endotracheal intubation is a life-sustaining procedure, its presence can deteriorate the structure and function of oropharynx, which may contribute to the difficulties in swallowing and subsequent oral intake. Estimated 62% of patients who had been intubated ≥48 hours will experience post-extubation dysphagia. Clearly, intervention is needed but studies are lacking in this regard. Thus, the objective of this pilot trial is to evaluate effects of an Oral Swallowing Care Program on swallowing and oral intake status in patients following prolonged endotracheal intubation.

This study employs a pre-and post-intervention design. The investigators were enrolled 63 post-extubated adult patients (50 years old and older) who had prolonged (≥48 hours) oral endotracheal intubation from six medical intensive care units at a medical center in Taipei, Taiwan.

Participants were assessed within 48 hours post-extubation for the baseline data, then a 14-day, daily Swallowing and Oral Care (SOC) Program involves toothbrushing/salivary gland massage, oral exercise(i.e., active/resistive range-of-motion[ROM] exercises for tongue, lips, and jaw), and advice on safe-swallowing strategies.

Outcome were assessed on 2nd, 7th, 14th, and 21st day post-extubation including oral health status, oral sensation (stereognosis, light touch and two-point discrimination), tongue and lip strength, salivary secretion, body weight. In addition, Three-Step Swallowing Screen (3-SSS) and Functional Oral Intake Scale(FOIS) were assessed daily. The data were analyzed by SPSS 12 software package.

ELIGIBILITY:
Inclusion criteria

* Adult patients (50 years old and older)
* People who had been extubated for over 48 hours and successfully extubated
* People or their legal representative who agree to participate in this study and sign the permit
* People who can communicate with Mandarin or Taiwanese

Exclusion criteria

* People who have diagnosis of neurological diseases such as cerebrovascular disease, Parkinson's disease or spinal injury, etc.
* People who have abnormal structure or function of oropharynx such as patients with head neck cancer or acquired/ inherited abnormal oropharynx structure
* People who currently have endotracheostomy
* People who are unconscious or have mental disability, having difficulty following the protocol or interacting with others
* People who are absolute quarantined. such as patients with open tuberculosis
* People who had swallowing difficulties before current intubation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Days to reach Oral intake status level 6 | 21 days post-extubation
  Using the "Functional Oral Intake Scale (FOIS)", a validated tool with established validity (81%-98%) and inter-rater reliabilities (0.86 to 0.91). The scale ranges from levels 1 to 7, level 1=Nothing by mouth; level 2=Tube dependent with minimal attempts of food or liquid; level 3=Tube dependent with consistent oral intake of food or liquid; level 4=Total oral diet of a single consistency; level 5=Total oral diet with multiple consistencies, but requiring special preparation or compensations; level 6=Total oral diet with multiple consistencies with special preparation, but with specific food limitations; level 7=Total oral diet with no restrictions.
whether return to total oral intake within 21 days post extubation | 21 days post-extubation
  Using the "Functional Oral Intake Scale (FOIS)", a validated tool with established validity (81%-98%) and inter-rater reliabilities (0.86 to 0.91). The scale ranges from levels 1 to 7, level 1=Nothing by mouth; level 2=Tube dependent with minimal attempts of food or liquid; level 3=Tube dependent with consistent oral intake of food or liquid; level 4=Total oral diet of a single consistency; level 5=Total oral diet with multiple consistencies, but requiring special preparation or compensations; level 6=Total oral diet with multiple consistencies with special preparation, but with specific food limitations; level 7=Total oral diet with no restrictions.
pass or fail Three-Step Swallowing Screen at 7th day post-extubation | on 7th day post-extubation
  Evaluation by using Three-Step Swallowing Screen(3-SSS). Participants were first assessed for prior history of dysphagia/feeding-tube dependence and signs of consciousness change, poor oxygen saturation (i.e., SaO2<90%; oxygen-mask dependence; reintubation), obvious drooling, or frequent choking on saliva. If negative, participants were then asked to swallow 3mL of water. If laryngeal elevation was identified with no signs of choking or wet voice, participants were asked to swallow 50mL of water; those without any signs of choking, wet voice, or slow swallowing were considered to pass the 3-SSS.
pass or fail Three-Step Swallowing Screen at 14th day post-extubation | on 14th day post-extubation
  Evaluation by using Three-Step Swallowing Screen(3-SSS). Participants were first assessed for prior history of dysphagia/feeding-tube dependence and signs of consciousness change, poor oxygen saturation (i.e., SaO2<90%; oxygen-mask dependence; reintubation), obvious drooling, or frequent choking on saliva. If negative, participants were then asked to swallow 3mL of water. If laryngeal elevation was identified with no signs of choking or wet voice, participants were asked to swallow 50mL of water; those without any signs of choking, wet voice, or slow swallowing were considered to pass the 3-SSS.
pass or fail Three-Step Swallowing Screen at 21st day post-extubation | on 21st day post-extubation
  Evaluation by using Three-Step Swallowing Screen(3-SSS). Participants were first assessed for prior history of dysphagia/feeding-tube dependence and signs of consciousness change, poor oxygen saturation (i.e., SaO2<90%; oxygen-mask dependence; reintubation), obvious drooling, or frequent choking on saliva. If negative, participants were then asked to swallow 3mL of water. If laryngeal elevation was identified with no signs of choking or wet voice, participants were asked to swallow 50mL of water; those without any signs of choking, wet voice, or slow swallowing were considered to pass the 3-SSS.

SECONDARY OUTCOMES:
Oral health status | on the 2nd, 7th and 14th day post-extubation
  The oral health status evaluated by Oral Assessment Guide(OAG), a validated tool with established validity and inter-rater reliabilities. The scores was coded as "1=no change", "2=moderate change", "3= severe change" of eight categories (voice, ability to swallow, lips, saliva, tongue, mucous membrane, gingiva, teeth). All scores are summed, ranges from 3 to 24.
Oral stereognosis | on the 2nd, 7th and 14th day post-extubation
  Oral stereognosis was measured by a set of five standardized researcher-made acrylic resin shapes (round, square, star, oval, and triangular), as suggested. Participants were given 30 s to visually inspect the test pieces along with the diagram of corresponding shapes before testing began.The variable are depicted in term of percentage of participants answered correct shape of each test piece (ranges 0~100%).
Oral light-touch sensation | on the 2nd, 7th and 14th day post-extubation
  Oral light touch sensation was measured with Semmes-Weinstein monofilaments. A standardized set of 5 monofilaments with values from 1.65 to 3.22 (log force) was used.
Oral two-point discrimination | on the 2nd, 7th and 14th day post-extubation
  The stereognostic ability of the tongue was tested using the MacKinnon-Dellon Disk-criminator. The variable are depicted in term of distance in millimeter (mm) when two-point sensation was perceived by participants.
Tongue and lip strength | on the 2nd, 7th, and 14th day post-extubation
  The tongue and lip strength assessed using the Iowa Oral Performance Instrument (IOPI System; IOPI Medical LLC, Carnation, WA, USA).
Salivary secretion | on the 2nd, 7th, and 14th day post-extubation
  Record salivary secretion using Modified Schirmer's test. With participants sitting upright, research nurses held a standardized 1-cm wide by 17-cm long Schirmer tear test strip vertically, with the rounded end of the strip placed at the floor of their mouth. At the end of 5 minutes, a wetting length in centimeter (cm) was recorded.
Body weight | on the 2nd, 7th, 14th and 21th day post-extubation.
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl CH Chen, Professor, Principal Investigator — Nursing Graduate Institute, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Solh A, Okada M, Bhat A, Pietrantoni C. Swallowing disorders post orotracheal intubation in the elderly. Intensive Care Med. 2003 Sep;29(9):1451-5. doi: 10.1007/s00134-003-1870-4. Epub 2003 Aug 2. PMID 12904855
- [Background] Macht M, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Postextubation dysphagia is persistent and associated with poor outcomes in survivors of critical illness. Crit Care. 2011;15(5):R231. doi: 10.1186/cc10472. Epub 2011 Sep 29. PMID 21958475
- [Background] Macht M, King CJ, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Post-extubation dysphagia is associated with longer hospitalization in survivors of critical illness with neurologic impairment. Crit Care. 2013 Jun 20;17(3):R119. doi: 10.1186/cc12791. PMID 23786755
- [Background] Kim MJ, Park YH, Park YS, Song YH. Associations Between Prolonged Intubation and Developing Post-extubation Dysphagia and Aspiration Pneumonia in Non-neurologic Critically Ill Patients. Ann Rehabil Med. 2015 Oct;39(5):763-71. doi: 10.5535/arm.2015.39.5.763. Epub 2015 Oct 26. PMID 26605174
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Tsai MH, Ku SC, Wang TG, Hsiao TY, Lee JJ, Chan DC, Huang GH, Chen CC. Swallowing dysfunction following endotracheal intubation: Age matters. Medicine (Baltimore). 2016 Jun;95(24):e3871. doi: 10.1097/MD.0000000000003871. PMID 27310972
- [Background] Brodsky MB, Huang M, Shanholtz C, Mendez-Tellez PA, Palmer JB, Colantuoni E, Needham DM. Recovery from Dysphagia Symptoms after Oral Endotracheal Intubation in Acute Respiratory Distress Syndrome Survivors. A 5-Year Longitudinal Study. Ann Am Thorac Soc. 2017 Mar;14(3):376-383. doi: 10.1513/AnnalsATS.201606-455OC. PMID 27983872
- [Background] Rassameehiran S, Klomjit S, Mankongpaisarnrung C, Rakvit A. Postextubation Dysphagia. Proc (Bayl Univ Med Cent). 2015 Jan;28(1):18-20. doi: 10.1080/08998280.2015.11929174. PMID 25552788
- [Background] Affoo RH, Trottier K, Garrick R, Mascarenhas T, Jang Y, Martin RE. The Effects of Tooth Brushing on Whole Salivary Flow Rate in Older Adults. Biomed Res Int. 2018 Feb 26;2018:3904139. doi: 10.1155/2018/3904139. eCollection 2018. PMID 29682540
- [Background] Park T, Kim Y. Effects of tongue pressing effortful swallow in older healthy individuals. Arch Gerontol Geriatr. 2016 Sep-Oct;66:127-33. doi: 10.1016/j.archger.2016.05.009. Epub 2016 Jun 3. PMID 27318884
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Lopez-Jornet P, Camacho-Alonso F, Bermejo-Fenoll A. A simple test for salivary gland hypofunction using Oral Schirmer's test. J Oral Pathol Med. 2006 Apr;35(4):244-8. doi: 10.1111/j.1600-0714.2006.00411.x. PMID 16519773
- [Background] Chen CC, Wu KH, Ku SC, Chan DC, Lee JJ, Wang TG, Hsiao TY. Bedside screen for oral cavity structure, salivary flow, and vocal production over the 14days following endotracheal extubation. J Crit Care. 2018 Jun;45:1-6. doi: 10.1016/j.jcrc.2017.11.035. Epub 2017 Dec 16. PMID 29257983
- [Background] Heffner JE. Swallowing complications after endotracheal extubation: moving from "whether" to "how". Chest. 2010 Mar;137(3):509-10. doi: 10.1378/chest.09-2477. No abstract available. PMID 20202944
- [Background] Su H, Hsiao TY, Ku SC, Wang TG, Lee JJ, Tzeng WC, Huang GH, Chen CC. Tongue weakness and somatosensory disturbance following oral endotracheal extubation. Dysphagia. 2015 Apr;30(2):188-95. doi: 10.1007/s00455-014-9594-x. Epub 2015 Feb 8. PMID 25663416
- [Background] Boliek CA, Rieger JM, Li SY, Mohamed Z, Kickham J, Amundsen K. Establishing a reliable protocol to measure tongue sensation. J Oral Rehabil. 2007 Jun;34(6):433-41. doi: 10.1111/j.1365-2842.2007.01735.x. PMID 17518978
- [Background] Rech RS, Baumgarten A, Colvara BC, Brochier CW, de Goulart B, Hugo FN, Hilgert JB. Association between oropharyngeal dysphagia, oral functionality, and oral sensorimotor alteration. Oral Dis. 2018 May;24(4):664-672. doi: 10.1111/odi.12809. Epub 2018 Feb 27. PMID 29164750
- [Derived] Wu CP, Xu YJ, Wang TG, Ku SC, Chan DC, Lee JJ, Wei YC, Hsiao TY, Chen CC. Effects of a swallowing and oral care intervention for patients following endotracheal extubation: a pre- and post-intervention study. Crit Care. 2019 Nov 9;23(1):350. doi: 10.1186/s13054-019-2623-2. PMID 31706360